CLINICAL TRIAL: NCT07160881
Title: Is There a More Affordable Method for Training in Cardiopulmonary Resuscitation - CPR? Comparing the Effectiveness of Standard CPR Manikins and CPR Pillows.
Brief Title: Effectiveness of CPR Pillow
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Aysegul Gunes, Health Science Faculty Lecturer (PhD. RN.), University of Beykent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: İstanbul Beykent Üniversitesi
Record Dates: First submitted 2025-08-20; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Healthy Participants
Keywords: basic life support; CPR; pillow maniquin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group using pillow maniquin (Experimental): This group will be given CPR training with a pillow manikin.
  Interventions: Behavioral: Pillow maniquin training

INTERVENTIONS:
Behavioral: Pillow maniquin training — In this initiative, participants will be trained with a low-cost mannequin in addition to standard training.

SUMMARY:
Pillows can be used to facilitate safe and effective learning and as a cheaper and more accessible alternative to manikins or computer-based methods for CPR training by non-healthcare professionals. The purpose of this study was to compare the effectiveness of pillows and manikins in CPR training.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age

Exclusion Criteria:

* No physical impairment is required to perform CPR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-09-17 (Estimated); Study Completion 2025-10-17 (Estimated)

PRIMARY OUTCOMES:
Cardiac compression number | 0. day (The parameter will be evaluated immediately after my ethics.)
  The number of compressions applied by the participants in one minute will be calculated.
Compression depth | 0. day (The parameter will be evaluated immediately after training.)
  Cardiac compression depth will be measured in cm.
Hand Position | 0. day (The parameter will be evaluated immediately after training.)
  The suitability of the compression area will be evaluated by the instructor.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Beykent University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No